CLINICAL TRIAL: NCT07352644
Title: Factors Affecting Attachment Loss in Clear Aligner Treatment: A Prospective Clinical Study
Brief Title: Factors Affecting Attachment Loss in Clear Aligner Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Şerife Şahin, Assistant Professor, Bezmialem Vakif University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022/19; 2022/19 (Other: Bezmialem Vakif University)
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Malocclusion; Crowded Teeth; Attachment
Keywords: ATTACHMENT; ATTACHMENT LOSS; c; CLEAR ALIGNER TREATMENT
MeSH Terms: conditions — Malocclusion; Crowding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clear Aligner Treatment (Experimental): Participants received clear aligner therapy (Invisalign®) with composite attachments bonded according to the manufacturer's protocol. Both conventional and optimized attachment types were used as part of the planned orthodontic treatment, and attachment loss was prospectively evaluated over a 6-month follow-up period.
  Interventions: Device: Clear Aligners with Composite Attachments

INTERVENTIONS:
Device: Clear Aligners with Composite Attachments — Participants received clear aligner therapy (Invisalign®, Align Technology, San Jose, CA, USA). Composite attachments were bonded according to the manufacturer's protocol using a high-viscosity composite. Both conventional and optimized attachment types were used as part of the planned orthodontic treatment, and attachment loss was prospectively evaluated during a 6-month follow-up period.

SUMMARY:
This prospective clinical study evaluated the incidence of composite attachment loss in patients undergoing clear aligner treatment and identified patient-, tooth-, and treatment-related factors associated with attachment debonding. Twenty-one patients were followed for six months, and attachment failures were recorded at routine visits. Outcomes were compared according to attachment type (conventional vs. optimized), attachment size, tooth type, dental arch, and patient-related factors.

DETAILED DESCRIPTION:
Composite attachments are integral to clear aligner therapy for improving force delivery, retention, and control of complex tooth movements. Despite their biomechanical importance, attachment loss remains a common clinical challenge and may compromise treatment efficiency and predictability. In this prospective study, attachments were bonded following the manufacturer's protocol using a high-viscosity composite. Patients were followed for six months, and attachment failures were documented with respect to type, size, tooth position, and patient-related behaviors. The primary objective was to determine the incidence of attachment loss and to identify factors associated with debonding, thereby contributing to clinical strategies that may reduce attachment failure and enhance treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

Permanent dentition. Mild to moderate crowding. No history of previous orthodontic treatment with fixed appliances or clear aligners

Exclusion Criteria:

Poor oral health. Bruxism. Crown restorations. Dental fluorosis. Enamel hypoplasia or other structural abnormalities affecting attachment bonding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Attachment Loss Rate | 6 months
  Proportion of composite attachments exhibiting complete detachment or partial debonding (irregular residual composite) during routine follow-up visits. Attachment loss was assessed by direct intraoral examination and tactile verification using a dental explorer.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No